CLINICAL TRIAL: NCT07149298
Title: Quality of Life In Patients With Allergic Conjunctivitis In Treatment With Sublingual Allergen Immunotherapy In A Referral Ophthalmological Hospital
Acronym: CVCA
Status: Active, not recruiting | Type: Observational
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Other Study IDs: CEI-2024/05/03; CB-013-2024 (Other: Instituto de Oftalmología Conde de Valenciana Comité de Bioseguridad); CI-014-2024 (Other: Instituto de Oftalmología Conde de Valenciana Comité de Investigación)
Record Dates: First submitted 2025-08-21; First posted 2025-08-29 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Allergic Conjunctivitis of Both Eyes
Keywords: Allergic Conjuntivitis; Allergy; Allergen; Life Quality; Allergen Immunotherapy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with conjunctivitis and treated with Sublingual Allergen Immunotherapy: 100 patients who attended the Conde de Valenciana Institute's Immunology Department from 2014 to 2023, diagnosed with conjunctivitis, treated with allergen-specific sublingual immunotherapy, completed all 10 vials of treatment, and completed at least eight quality-of-life questionnaires.

SUMMARY:
The goal of this observational study is to evaluate both clinical changes and quality-of-life outcomes in patients with allergic conjunctivitis treated with allergen-specific immunotherapy, integrating objective clinical parameters and validated quality-of-life measures to obtain a comprehensive view of the therapeutic impact.

DETAILED DESCRIPTION:
BACKGROUND: Allergic conjunctivitis (AC) is an inflammatory disease of the ocular surface that may be affecting people's quality of life. Studies have shown that allergic diseases are a risk factor for depression, sleep problems, and affect the patient's mood. Allergen-specific sublingual immunotherapy has been shown to be beneficial for the treatment of asthma and allergic rhinitis.

JUSTIFICATION: There are no studies demonstrating whether allergen-specific sublingual immunotherapy improves the different dimensions of quality of life affected by allergic conjunctivitis.

HYPOTHESIS: Quality of life in allergic conjunctivitis will improve with the administration of allergen-specific sublingual immunotherapy.

GENERAL OBJECTIVE: To define changes in quality of life in patients with allergic conjunctivitis before, during, and after allergen-specific sublingual immunotherapy using a standardized quality of life questionnaire at an ophthalmology referral hospital.

MATERIAL AND METHODS: A retrospective, observational, and longitudinal study will be conducted, reviewing 100 patient records of patients who attended the Immunology Department of the Conde de Valenciana Institute from 2018 to 2023, diagnosed with conjunctivitis, treated with allergen-specific sublingual immunotherapy, completed all 3 years of treatment, and completed at least 8 quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patient records containing complete information
* Both sexes
* Age range: 6 to 86 years
* Between 2018 and 2023
* Diagnosed with allergic conjunctivitis
* Who have received treatment with allergen-specific sublingual immunotherapy
* With 8 assessments from the immunology and cornea department
* With 7 quality of life questionnaires completed by the patient

Exclusion Criteria:

* Patient records for other inflammatory ocular conditions
* Those with chronic diseases
* Those who have received naturopathic or immunomodulatory treatment during the follow-up period for allergen-specific sublingual immunotherapy

Ages: 6 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 100 patients who attended the Conde de Valenciana Institute's Immunology Department from 2018 to 2023, diagnosed with conjunctivitis, treated with allergen-specific sublingual immunotherapy, completed 3 years of treatment, and completed at least eight quality-of-life questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-03-24 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Quality of life evaluated by the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Spanish version for Mexico in patients with Allergic Conjunctivitis treated with sublingual allergen immunotherapy. | Before Sublingual Immunotherapy
  To evaluate the quality of life in patients with Allergic Conjunctivitis treated with sublingual allergen immunotherapy using the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Spanish version for Mexico. This questionnaire features 28 items grouped in 7 domains: activities, sleep, other symptoms, practical problems, nasal symptoms, eye symptoms, emotional. For each item, the minimum score is 0 and the maximum score is 6. After the questionnaire is completed, a mean score is calculated. A higher overall score indicates a poorer quality of life.
Quality of life in patients with Allergic Conjunctivitis treated with sublingual allergen immunotherapy evaluated using the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Spanish version for Mexico. | From enrollment to the end of the 6th month of Allergen Immunotherapy treatment
  To evaluate the quality of life in patients with Allergic Conjunctivitis during 6 months of sublingual allergen immunotherapy using the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Spanish version for Mexico. This questionnaire features 28 items grouped in 7 domains: activities, sleep, other symptoms, practical problems, nasal symptoms, eye symptoms, emotional. For each item, the minimum score is 0 and the maximum score is 6. After the questionnaire is completed, a mean score is calculated. A higher overall score indicates a poorer quality of life.
Quality of life in patients with Allergic Conjunctivitis treated with sublingual allergen immunotherapy using Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Spanish version for Mexico. | From enrollment until 3 years of treatment with sublingual immunotherapy
  To evaluate quality of life in patients with Allergic Conjunctivitis after completing allergen-specific sublingual immunotherapy using the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Spanish version for Mexico. This questionnaire features 28 items grouped in 7 domains: activities, sleep, other symptoms, practical problems, nasal symptoms, eye symptoms, emotional. For each item, the minimum score is 0 and the maximum score is 6. After the questionnaire is completed, a mean score is calculated. A higher overall score indicates a poorer quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Oftalmología FAP Conde de Valenciana, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
As Supplementary Material in the publication
Supporting Information: Study Protocol
Time Frame: After publication
Access Criteria: The information will be completely public.

REFERENCES:
- [Background] Sanchez-Hernandez MC, Montero J, Rondon C, Benitez del Castillo JM, Velazquez E, Herreras JM, Fernandez-Parra B, Merayo-Lloves J, Del Cuvillo A, Vega F, Valero A, Panizo C, Montoro J, Matheu V, Lluch-Bernal M, Gonzalez ML, Gonzalez R, Dordal MT, Davila I, Colas C, Campo P, Anton E, Navarro A; SEAIC 2010 Rhinoconjunctivitis Committee; Spanish Group Ocular Surface-GESOC. Consensus document on allergic conjunctivitis (DECA). J Investig Allergol Clin Immunol. 2015;25(2):94-106. PMID 25997302
- [Background] Devillier P, Dreyfus JF, Demoly P, Calderon MA. A meta-analysis of sublingual allergen immunotherapy and pharmacotherapy in pollen-induced seasonal allergic rhinoconjunctivitis. BMC Med. 2014 May 1;12:71. doi: 10.1186/1741-7015-12-71. PMID 24885894
- [Background] Calderon-Ezquerro, M. C., Guerrero-Guerra, C., Galán, C., Serrano-Silva, N., Guidos-Fogelbach, G., Jiménez-Martínez, M. C., Larenas-Linnemann, D., López Espinosa, E. D., & Ayala-Balboa, J. (2018). Pollen in the atmosphere of Mexico City and its impact on the health of the pediatric population. Atmospheric Environment (Oxford, England: 1994), 186, 198-208. https://doi.org/10.1016/j.atmosenv.2018.05.006
- [Background] Barrón-Campos, A., Velázquez-Samano, G., Velasco-Medina, A., Barrón-Soto, M. (2024). Evaluación de la calidad de vida de pacientes con rinitis alérgica por medio del cuestionario Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ). Anales de Otorrinolaringología Mexicana 69:4. https://doi.org/10.24245/aorl.v69i4.10165